CLINICAL TRIAL: NCT00553527
Title: Biomet Humeral Stem Data Collection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to terminate the project due to low multi-center enrollment.
Sponsor: Vanderbilt University (Other)
Responsible Party: Dr. Donald Lee, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 070144
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Humeral Stem Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Patient will receive standard of care humeral stem replacement. Only a data collection study. There will be no changes in standard of care for diagnosis.
  Interventions: Procedure: Humeral Stem replacement surgery

INTERVENTIONS:
Procedure: Humeral Stem replacement surgery — Patient will receive humeral stem replacement.

SUMMARY:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of Biomet Humeral Stems.

DETAILED DESCRIPTION:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of Biomet Humeral Stems.

All stems on which data will be collected are legally marketed and none of the devices are investigational or experimental. This data collection effort will document the clinical outcomes of the humeral stems. The data gathered will be collated and used to provide feedback to designing engineers, support marketing efforts, and answer potential questions from reimbursement agencies.

Inclusion/Exclusion criteria are within the indications and contraindications stated in the labeling, cleared by the FDA, for the device. Surgical techniques and patient care are to be standard for the surgeon participating in the protocol. There will be no experimental or investigational surgical techniques used. The devices and products are to be used in accordance with their instructions for use and/or approved labeling.

The outcomes and data collected include:

UCLA End-Result Score Radiographic Evaluation

Survivorship will be documented by asking the surgeon to record revisions, complications, and device related events.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid Arthritis
* Correction of functional deformity
* Patient selection factors to be considered:

  1. Need to obtain pain relief and improve function
  2. Ability and willingness of the patient to follow instructions, including control of weight and activity levels
  3. A good nutritional state of the patient
  4. The patient must have reached full skeletal maturity

Exclusion Criteria:

* Patients who have infection, sepsis, and osteomyelitis
* Patients who are uncooperative or have neurologic disorders who is capable or unwilling to follow directions
* Patients who have osteoporosis
* Patients who have metabolic disorders which may impair bone function
* Patients with osteomalacia
* Patients with distant foci of infections which may spread to the implant site
* Patients with rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Patients who are pregnant
* Patients who are under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The outcome will be measured using the data collection sheets collected at each follow-up visit. | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Lee, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Hand Center, Nashville, Tennessee, United States